CLINICAL TRIAL: NCT05174793
Title: Urine Color Expressed in CIE L*a*b* Colorspace During Rapid Changes in Hydration Status
Brief Title: Using Urine Color as a Marker of Hydration Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Michael J. Buono, Professor, San Diego State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ENS1; 0146 (Other: SDSU IRB)
Record Dates: First submitted 2021-11-22; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration | interventions — Fluid Therapy

STUDY DESIGN:
Intervention Model Description: urine color was measured during dehydration and rehydration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dehydration to rehydration (Experimental): subjects were rehydrated following 2% dehydration
  Interventions: Other: dehydration and rehydration
- euhydration to dehydration (Experimental): subjects were dehydrated by 2% with exercise in the heat
  Interventions: Other: dehydration and rehydration

INTERVENTIONS:
Other: dehydration and rehydration — dehydration and rehydration

SUMMARY:
The purpose of this study was to determine if rapid changes in hydration status could be determined by urine color expressed in CIE color space

DETAILED DESCRIPTION:
The study will examine if urine color expressed in CIE color space can reflect hydration status. Hydration staus will be rapidly altered via exercise in the heat.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age,
* no previous heat intolerance

Exclusion Criteria:

- Pregnant women,

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
can urine color expressed in CIE color space reflect hydration status | one hour dehydration and rehydration
  urine color expressed in CIE color space

CONTACTS AND LOCATIONS:
Overall Officials: Michael Buono, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT05174793/Prot_SAP_000.pdf